CLINICAL TRIAL: NCT03435718
Title: An Assessor Blind, Randomized, Comparative Study of the Efficacy of Different Doses of Oxfendazole Compared to Single Dose Albendazole in the Treatment of Trichuris Trichiura Infection in Adults
Brief Title: Efficacy of Oxfendazole in the Treatment of Trichuris Trichiura Infection in Adults
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oxfendazole Development Group (Other)
Collaborators: Universidad Peruana Cayetano Heredia, Lima, Peru (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXF2 v3.21
Record Dates: First submitted 2018-02-02; First posted 2018-02-19 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Trichuris Infection
Keywords: oxfendazole; albendazole; Trichuris trichiura
MeSH Terms: conditions — Trichuriasis | interventions — oxfendazole; Albendazole

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a field trial. Patients will be randomly assigned to one of five treatment groups: 6 mg/kg, 15 mg/kg or 30 mg/kg oxfendazole as a single dose; 15 mg/kg oxfendazole on three consecutive days; or 400 mg albendazole as a single dose (50 patients per group). The main objective of this study is to assess the efficacy (Cure Rate) of oral oxfendazole. Secondary objectives are to assess the Egg Reduction Rate for Trichuris in those subjects not cured of infection, to assess the efficacy (Cure Rate and Egg Reduction Rate) of oxfendazole against other common intestinal helminth infections, and to assess the safety and tolerability of oxfendazole treatment in adult patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each patient's treatment condition will be masked by a code assigned at randomization. The study pharmacist will know this assignment. A person other than the investigator will administer the drug as directed by the pharmacists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- OXF6 (Experimental): Patients receive a single 6 mg/kg dose of oxfendazole administered orally.
  Interventions: Drug: Oxfendazole
- OXF15 (Experimental): Patients receive a single 15 mg/kg dose of oxfendazole administered orally.
  Interventions: Drug: Oxfendazole
- OXF30 (Experimental): Patients receive a single 30 mg/kg dose of oxfendazole administered orally.
  Interventions: Drug: Oxfendazole
- OXF15x3 (Experimental): Patients receive a 15 mg/kg dose of oxfendazole administered orally once a day for each of three consecutive days.
  Interventions: Drug: Oxfendazole
- ALB400 (Active Comparator): Patients receive a single 400 mg/kg dose of albendazole administered orally.
  Interventions: Drug: Albendazole

INTERVENTIONS:
Drug: Oxfendazole — oral suspension
  Arms: OXF15; OXF15x3; OXF30; OXF6
Drug: Albendazole — tablet
  Arms: ALB400

SUMMARY:
The main objective of this study is to provide data on the efficacy profile of different doses of oxfendazole when used in Trichuris trichiura infection. The drug will be also be examined for efficacy against other common nematodes encountered in man (Ascaris lumbricoides, Ancylostoma duodenale, Necator americanus). The study will also provide data on the safety and tolerability of the oxfendazole in patients.

DETAILED DESCRIPTION:
This is an assessor blind, randomized, comparative study in adult patients with proven intestinal infection with Trichuris trichiura to be conducted as a field study. Patients meeting the study entry criteria will receive either 6 mg/kg or 15 mg/kg or 30 mg/kg of oxfendazole as a single oral dose, three single doses of oxfendazole on consecutive days, or albendazole 400mg as a single oral dose. Stool samples will be obtained and examined prior to treatment and at 7, 14 and 21 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatient, more than 18 years and less than 65 years of age.
2. Written or witnessed oral informed consent has been obtained.
3. Trichuris trichiura demonstrated in stool samples obtained during the week before enrolment: The presence of Ascaris lumbricoides, Necator americanus, Ancylostoma duodenalis or other helminths will not be a cause for exclusion.
4. Willingness to comply with the requirements of the protocol and particularly to provide 4 stool samples, pretreatment and 7, 14 and 21 days after treatment.
5. Female patients of child bearing potential, who are using an established method of birth control (surgically sterile, intra-uterine contraceptive device, oral contraceptives, diaphragm in combination with contraceptive cream or foam, or condom in combination with contraceptive cream or foam) may be included

Exclusion Criteria:

1. The patient has demonstrated a previous hypersensitivity reaction to benzimidazole or other related compound.
2. Presence of other helminths without Trichuris trichiura. Non-target species may be present and details of response will be recorded.
3. The patient has diarrhoeal disease that would interfere with the evaluation of stool samples.
4. The patient has received an anthelminthic in the 2 weeks prior to enrolment into the study.
5. The patient has received an investigational drug within 30 days or 5 half-lives (whichever is longer) of the screening visit or is scheduled to receive such a drug during the study period.
6. The patient has a concomitant infection or any other underlying disease that would compromise the diagnosis and the evaluation of the response to the study medication.
7. The patient has a known history of renal dysfunction or plasma creatinine ≥ 1.5 times upper limit of normal for age or a known history of hepatic dysfunction or liver enzymes ≥ 1.5 times upper limit of normal.
8. The patient is a female who is pregnant, lactating or planning a pregnancy during the study, or is not practicing any form of contraception (see inclusion criteria (4.2.5).
9. The patient is unwilling or unable to take part in this study.
10. The patient has previously been enrolled in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
cure d14 | Day 14 of follow up
  absence of eggs of Trichuris trichiura (determined by the Kato Katz method) in stool samples of treated patients
cure d7 | Day 7 of follow up
  absence of eggs of Trichuris trichiura (determined by the Kato Katz method) in stool samples of treated patients

SECONDARY OUTCOMES:
improvement d21 | Day 21 of follow up
  reduction (with respect to the baseline count of that individual) in number of eggs of Trichuris trichiura (determined by the Kato Katz method) in stool samples of treated patients
improvement d14 | Day 14 of follow up
  reduction (with respect to the baseline count of that individual) in number of eggs of Trichuris trichiura (determined by the Kato Katz method) in stool samples of treated patients
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0, d7 | Day 7 of follow up
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0, d14 | Day 14 of follow up
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0, d21 | Day 21 of follow up
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Héctor Hugo Garcia, MD PhD, Principal Investigator — Oxfendazole Development Group

IPD SHARING:
Plan to Share IPD: Undecided
The data will be uploaded to the clinicaltrials.gov website, and a publication will be prepared